CLINICAL TRIAL: NCT05948397
Title: To Use the Combined Version of ICIQ-SF and Quality of Life Scale in Mixed Urinary Incontinence
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Ersin Köseoglu, MD, Koç University
Other Study IDs: KocUrol2
Record Dates: First submitted 2023-07-09; First posted 2023-07-17 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Incontinence, Urge; Incontinence Stress; Quality of Life
MeSH Terms: conditions — Urinary Incontinence, Urge; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Female patients admitted to urology outpatient clinic with mixed urinary incontinence.
  Interventions: Diagnostic Test: Combined version of International Consultation on Incontinence Questionnaire Short Form (ICIQ SF) and quality of life scale; Diagnostic Test: Bladder diary; Diagnostic Test: Pad test

INTERVENTIONS:
Diagnostic Test: Combined version of International Consultation on Incontinence Questionnaire Short Form (ICIQ SF) and quality of life scale — A combined version of International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) and quality of life scale would be given to all patients. The sum of the responses for the third, fourth and fifth questions and quality of life scale scores will be recorded.
Diagnostic Test: Bladder diary — Bladder diary is an online application. Frequency, nocturia, functional bladder capacities will be reported. More than 8 urination during daytime will be recorded as overactive bladder. More than 1 interruption of sleep for urination at night is nocturia. Functional bladder capacity below 100 ml will be defined as decreased bladder capacity, while capacity over 400 ml will be reported as increased bladder capacity and compliance
Diagnostic Test: Pad test — One-hour pad test.
  * the test is started by putting one pre-weighted pad without patient voiding, -patient drinks 500 ml of sodium-free liquid in <15 min- then sits or rests,
  * patient walks for 30 min, including climbing one flight of stairs (up and down),
  * patient performs the following activities: standing up from sitting (10 ), coughing vigorously (10 ), running on the spot for 1 min, bending to pick up an object from the floor (5 ), and washing hands in running water for 1 min (this activity program may be modified according to the patient's physical fitness),
  * the total amount of urine leaked is determined by weighing the pad. In the analysis of 1-hr pad test, an increase of 1-10 g is classified as representing mild incontinence, 11-50 g moderate and >50 g severe incontinence. The values for 24-hr pad test are classified as follows: Mild (4-20 g/ 24 hr), moderate (21-74 g/24 hr), and severe (>75 g/24 hr) incontinence

SUMMARY:
The goal of this observational study is detecting the dominant component of mixed urinary incontinence via a combined version of ICIQ-SF and quality of life scale. The main question it aims to answer is:

1. Which component (urgency or stress) urinary incontinence bothers the patient more?

DETAILED DESCRIPTION:
Female patients with mixed urinary incontinence will be given a combined version of ICIQ-SF and quality of life scale on the first visit. Additionally, a bladder diary and 1-hour pad test will be performed on the same visit. After deciding the appropriate treatment, on the 1-month visit (second visit) the same tests will be repeated and scores will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Female patients above 18 years old with mixed urinary incontinence

Exclusion Criteria:

* Non-Turkish speakers
* Poor conscious level
* Immobile patients

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients above 18 years old.
Study Population: Females with mixed urinary incontinence
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire Short Form | 1 month
  Questionnaire
Pad test | 1 month
  Diagnostic Test
Bladder diary | 1 month
  Diagnostic Test

IPD SHARING:
Plan to Share IPD: No